CLINICAL TRIAL: NCT06243406
Title: Study on the Biomarkers to Predict the Response to Anti-vascular Endothelial Growth Factor Treatment for Choroidal Neovascularization
Brief Title: Study on the Biomarkers of Anti-VEGF Treatment for Choroidal Neovascularization
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: BJ-2022-012
Record Dates: First submitted 2024-01-29; First posted 2024-02-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intravitreal injection of anti-VEGF — Intravitreal injection of anti- vascular endothelial growth factor (VEGF) treatment

SUMMARY:
Choroidal neovascularization (CNV), also known as subretinal neovascularization, is a proliferative change from choroidal capillaries that has become one of the most important causes of blindness worldwide. CNV can occur in a variety of fundus diseases, including pathologic myopia, polypoidal choroidal vasculopathy. At present, intravitreal injection of anti-vascular endothelial growth factor (VEGF) drugs is the first-line effective treatment for CNV. Although a number of clinical studies have shown that the treatment of CNV with anti-VEGF drugs has achieved good visual and anatomical effects, there are still some patients whose CNV has not decreased significantly or even progressed continuously after treatment. Rapid advances in imaging technology have made it possible to explore the quantitative and qualitative characteristics of choroid and CNV, especially swept source optical coherence tomography angiography (SS-OCTA).

The objectives are to improve the OCTA typing of CNV and analyze the vascular morphological characteristics of each type; to identify the changes in vascular characteristics of CNV after anti-VEGF treatment in vitreous cavity; and to elucidate the predictive effects of neovascularization and choroidal vascular characteristics on visual acuity and anatomic effects of vitreous anti-VEGF drug treatment for CNV.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Active choroidal neovascularization (activity criteria: blood vessel leakage confirmed by FFA, or subretinal fluid accumulation or bleeding seen by OCT)
* History of anti-VEGF drug therapy
* At least 3 months of follow-up data.

Exclusion Criteria:

* Unable to complete the examination due to severe cataract or vitreous hemorrhage
* Any retinal diseases except choroidal neovascularization, such as multifocal choroiditis, diabetic retinopathy
* History of intraocular surgery

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with choroidal neovascularization, who received standard 3-monthly anti-VEGF treatment.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
choroidal thickness | 3 months
  central choroidal thickness measured by SS-OCTA
Central retinal thickness | 3 months
  central retinal thickness changes measured by SS-OCTA
Best-corrected visual acuity | 3 months
  Best-corrected visual acuity changes from baseline to 3 months

SECONDARY OUTCOMES:
choroidal vascularity index | 3 months
  the ratio of vascular area to the total choroidal area measured by SS-OCTA

IPD SHARING:
Plan to Share IPD: No